CLINICAL TRIAL: NCT03076619
Title: A Clinical Study of Fundus Findings in Toxaemia of Pregnancy (Pregnancy Induced Hypertension)
Brief Title: A Clinical Study of Fundus Findings in Toxaemia of Pregnancy
Status: Completed | Type: Observational
Sponsor: B. J. Medical College, Ahmedabad (Other Government)
Collaborators: M and J Western Regional Institute of Ophthalmology,Ahmedabad. (Unknown)
Responsible Party: Principal Investigator, Dr.Rahul Navinchandra Bakhda MS., Consultant Ophthalmologist, Ex-Resident, M and J Western Regional Institute of Ophthalmology, B. J. Medical College, Ahmedabad
Other Study IDs: Postgraduation Thesis; DRKS00011324 (Registry Identifier: The German Clinical Trials Register -Deutsche Register Klinischer Studien); ChiCTR-OOC-16010171 (Registry Identifier: Chinese Clinical Trial Registry-ChiCTR); UMIN000024722 (Registry Identifier: UMIN Clinical Trials Registry (UMIN-CTR)); U1111-1189-6165 (Registry Identifier: International Clinical Trials Registry Platform (ICTRP)); TCTR20161221005 (Registry Identifier: Thai Clinical Trials Registry (TCTR))
Record Dates: First submitted 2016-10-30; First posted 2017-03-10 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: pregnancy induced hypertension; ophthalmoscopy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical ophthalmoscopy in PIH: An observational study in which the patients for the study are selected from antenatal clinic, antenatal ward and "preeclampsia and eclampsia room" in Department of Obstetrics and Gynecology and general ophthalmic OPD in case of ambulatory patients during the period of November 2003 to June 2006 randomly.
  Interventions: Other: clinical ophthalmoscopy

INTERVENTIONS:
Other: clinical ophthalmoscopy — To study the role of clinical ophthalmoscopy in PIH in diagnosis, prognosis, differential diagnosis, line of treatment and effect of treatment.

SUMMARY:
Toxemia of pregnancy is a recognized entity for over 2000 years with its known complications and fatality. Nowadays, a most accepted terminology for the following defined syndrome is "hypertensive disorders in pregnancy" given by American College of Obstetrics and Gynecology. It is an important cause of maternal and fetal morbidity and mortality. Pregnancy induced hypertension (PIH) was classified as gestational hypertension, preeclampsia, severe preeclampsia and eclampsia. PIH is a hypertensive disorder in pregnancy that occurs after 20 weeks of pregnancy in the absence of other causes of elevated blood pressure (BP) (BP >140/90 mmHg measured two times with at least of 4 hour interval) in combination with generalized edema and/or proteinuria (>300 mg per 24 hrs). When there is significant proteinuria it is termed as preeclampsia; seizure or coma as a consequence of PIH is termed as eclampsia. Preeclampsia was classified into mild and severe preeclampsia.

Mild eclampsia-BP >140/90 mmHg, proteinuria+, and/or mild edema of legs, Severe preeclampsia-BP >160/110 mmHg,proteinuria++ or ++++, headache, cerebral or visual disturbances, epigastric pain, impaired liver function tests and increase in serum creatinine.

Proteinuria was tested using dipstick method as +=0.3 gm/L, ++=1 gm/L, and +++=3 gm/L.

The pathological changes of this disease appear to be related to vascular endothelial dysfunction and its consequences (generalized vasospasm and capillary leak). Ocular involvement is common in PIH.Common symptoms are blurring of vision, photopsia, scotomas and diplopia. Visual symptoms may be the precursor of seizures.Progression of retinal changes correlates with progression of PIH and also with the fetal mortality due to similar vascular ischemic changes in placenta.Vasospastic manifestations are reversible and the retinal vessels rapidly return to normal after delivery. Ophthalmoscope should be rated next to the sphygmomanometer as an instrument of diagnostic importance in cases of PIH. Ophthalmoscopy does not only helps in diagnosing the disease but repeated observations assist in assessing the severity, progress of disease, response to treatment if any and ultimate outcome or prognosis.

DETAILED DESCRIPTION:
An observational study in which the patients for the study are selected from antenatal clinic, antenatal ward and "preeclampsia and eclampsia room" in Department of Obstetrics and Gynecology and general Ophthalmic Out Patient Department(OPD) in case of ambulatory patients during the period of November 2003 to June 2006 randomly.In every case, detail obstetric history including a detail antenatal history was taken. General examination and relevant pathological investigations like routine blood count, HIV, HBsAg, renal function tests, TORCH complex etc., were carried out. In every case, pupil was dilated with homatropine (2%) eye drops. Then detailed ophthalmic examination was carried out with special emphasis on direct ophthalmoscopy apart from visual acuity of both eyes and anterior segment examination. Fundus findings were noted in detail, changes in the color of the disc, disc margin, physiological cup, changes in retinal blood vessels especially caliber of vessels, arterio-venous (AV) ratio,changes in vessel wall, blood column, appearance of vascular light reflex, changes at AV crossings, changes in macular area and changes in background, overall appearance, presence of hemorrhages, exudates or any pathology were recorded.

Fundus changes were graded as per modified Keith, Wagner and Barker classification.Assessment of prognosis as regards to vision and life (mortality) was made.

ELIGIBILITY:
Inclusion Criteria:

* Cases of Pregnancy Induced Hypertension.

Exclusion Criteria:

* Cases complicated by malignancy, renal, liver or other secondary manifestations.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: An observational study in which the patients for the study are selected from antenatal clinic, antenatal ward and "preeclampsia and eclampsia room" in Department of Obstetrics and Gynecology and general ophthalmic OPD in case of ambulatory patients during the period of November 2003 to June 2006 randomly.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2003-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The relation of positive fundus changes with number of cases of pregnancy induced hypertension | Nov. 2003 to June 2006 randomly
  Correlation of fundus changes with disease entity.In every case detail obstetric history, general examination and relevant pathological investigations were carried out. In every case, pupil was dilated with homatropine (2%) eye drops and detailed ophthalmic examination was carried out.
The relation of number of cases of PIH and positive fundus findings with number of gravida | Nov. 2003 to June 2006 randomly
  Correlation of fundus changes with gravida.
Relationship between total number of cases of PIH and fundus changes according to age | Nov. 2003 to June 2006 randomly
  Correlation of fundus changes with age.
Relationship between number of cases of PIH and fundus changes according to duration of pregnancy | Nov. 2003 to June 2006 randomly
  Correlation of fundus changes with duration of pregnancy
The relation of number of cases of PIH and fundus findings with systolic blood pressure | Nov. 2003 to June 2006 randomly
  In every case detail obstetric history, general examination and relevant pathological investigations were carried out. In every case, pupil was dilated with homatropine (2%) eye drops and detailed ophthalmic examination was carried out.
  Fundus findings were noted in detail.
The relation of number of cases of PIH and fundus findings with diastolic blood pressure | Nov. 2003 to June 2006 randomly
  In every case detail obstetric history, general examination and relevant pathological investigations were carried out. In every case, pupil was dilated with homatropine (2%) eye drops and detailed ophthalmic examination was carried out.
  Fundus findings were noted in detail.
The relation of number of cases of PIH according to fundus changes (according to modified Keith, Wagner and Barker classification) | Nov. 2003 to June 2006 randomly
  In every case detail obstetric history, general examination and relevant pathological investigations were carried out. In every case, pupil was dilated with homatropine (2%) eye drops and detailed ophthalmic examination was carried out.
  Fundus findings were noted in detail.
The relation of individual fundus findings with no. of cases of PIH | Nov. 2003 to June 2006 randomly
  Significance of individual fundus changes were noted

SECONDARY OUTCOMES:
Distribution of PIH cases on fetal outcome | Nov. 2003 to June 2006 randomly
  Assessment of prognosis as regards to vision and life (mortality) was made.i.e correlation of fundus changes with fetal outcome.
The relation of fundus changes with perinatal mortality | Nov. 2003 to June 2006 randomly
  Assessment of prognosis as regards to vision and life (mortality) was made.i.e correlation of fundus changes with fetal outcome and perinatal mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Rahul Bakhda, M.S., Principal Investigator — Ex-Resident,M and J Western Regional Institute of Ophthalmology, B.J.Medical College and Civil Hospital Campus, Ahmedabad-380016.Gujarat. 07922680360 07922680314 Fax:07922680360
Locations (1):
- M and J Western Regional Institute of Ophthalmology, B.J.Medical College and Civil Hospital Campus, Ahmedabad-380016.Gujarat. 07922680360 07922680314 Fax:07922680360, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakhda RN. Clinical study of fundus findings in pregnancy induced hypertension. J Family Med Prim Care. 2016 Apr-Jun;5(2):424-429. doi: 10.4103/2249-4863.192364. PMID 27843854
- See also: Published article — http://www.jfmpc.com/article.asp?issn=2249-4863;year=2016;volume=5;issue=2;spage=424;epage=429;aulast=Bakhda